CLINICAL TRIAL: NCT03262675
Title: National Tunisian Registry of Heart Failure
Acronym: NATURE-HF
Status: Completed | Type: Observational
Sponsor: Dacima Consulting (Other)
Collaborators: Société Tunisienne de Cardiologie & de Chirurgie Cardio-Vasculaire (Unknown)
Responsible Party: Sponsor
Other Study IDs: DAC-002-NATUREHF
Record Dates: First submitted 2017-08-22; First posted 2017-08-25 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Heart Failure
Keywords: Heart Failure; Acute Heart Failure; Chronic Heat Failure; Cardiovascular diseases; Heart diseases; Registry; Tunisia
MeSH Terms: conditions — Heart Failure; Cardiovascular Diseases; Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
NATURE-HF is an observational, multicentric and longitudinal study of heart failure performed with 100 tunisian cardiologists.

DETAILED DESCRIPTION:
The NATURE-HF is a national clinical non-interventional registry of heart failure, carried out in Tunisia at cardiology departments in hospitals and in liberal cardiology consultations. 100 cardiologists participate in the enrollment of the eligible patients as investigators. A Committee of Experts validates the protocol methodology and supervises the data-management. A Steering Committee helps investigators to monitor their patient inclusions, performs audit trails and prepares the statistical analysis plan for the study.

Collected data are managed by the DACIMA Clinical Suite®, the electronic data capture platform which complies with the FDA 21 CFR part 11 requirements (Food and Drug Administration 21 Code of Federal Regulations part 11), the HIPAA specifications (Health Insurance Portability and Accountability Act), and the ICH standards (International Conference on Harmonisation).

ELIGIBILITY:
Inclusion Criteria:

* Patient with chronic heart failure
* Patient with acute heart failure (new onset or not)
* The diagnosis of heart failure is at the discretion of the investigator
* Informed and signed consent

Exclusion Criteria:

* Life expectancy <12 months for extra cardiac disease
* Isolated Right Heart Failure
* Pregnant woman
* Renal failure with creatinine clearance < 15 ml / min
* Hemodialysis patients
* Cardiac surgery planned within 3 months
* Congenital heart disease

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with heart failure
Sampling Method: Non-Probability Sample
Enrollment: 2040 (Actual)
Dates: Start 2017-10-16 (Actual); Primary Completion 2017-11-22 (Actual); Study Completion 2019-01-12 (Actual)

PRIMARY OUTCOMES:
Cardiovascular death | Time-To-Event measure up to 12 months from baseline
  Incidence of cardiovascular death including sudden death, death from refractory heart failure and death from stroke

SECONDARY OUTCOMES:
Heart Failure Readmission | At 1, 3 and 12 months from patient enrollment
  Incidence of heart failure readmissions
Global Death | Time-To-Event measure up to 12 months from baseline
  Incidence of death of all causes (cardiovascular death and non-cardiovascular death)

CONTACTS AND LOCATIONS:
Overall Officials: Faouzi Addad, Professor, Study Chair — Société Tunisienne de Cardiologie et de Chirurgie Cardiovasculaire
Locations (1):
- Société Tunisienne de Cardiologie & de Chirurgie Cardio-Vasculaire, Tunis, Tunisie, Tunisia

IPD SHARING:
Plan to Share IPD: Yes
Clinical Study Report
Supporting Information: CSR
Time Frame: Already available
Access Criteria: Free access
URL: http://www.stcccv-tunisie.com/files/RegistreNatureHF_SFC2019.pdf

REFERENCES:
- [Derived] Abid L, Kammoun I, Ben Halima M, Charfeddine S, Ben Slima H, Drissa M, Mzoughi K, Mbarek D, Riahi L, Antit S, Ben Halima A, Ouechtati W, Allouche E, Mechri M, Yousfi C, Khorchani A, Abid O, Sammoud K, Ezzaouia K, Gtif I, Ouali S, Triki F, Hamdi S, Boudiche S, Chebbi M, Hentati M, Farah A, Triki H, Ghardallou H, Raddaoui H, Zayed S, Azaiez F, Omri F, Zouari A, Ben Ali Z, Najjar A, Thabet H, Chaker M, Mohamed S, Chouaieb M, Ben Jemaa A, Tangour H, Kammoun Y, Bouhlel M, Azaiez S, Letaief R, Maskhi S, Amri A, Naanaa H, Othmani R, Chahbani I, Zargouni H, Abid S, Ayari M, Ben Ameur I, Gasmi A, Ben Halima N, Haouala H, Boughzela E, Zakhama L, Ben Youssef S, Nasraoui W, Boujnah MR, Barakett N, Kraiem S, Drissa H, Ben Khalfallah A, Gamra H, Kachboura S, Bezdah L, Baccar H, Milouchi S, Sdiri W, Ben Omrane S, Abdesselem S, Kanoun A, Hezbri K, Zannad F, Mebazaa A, Kammoun S, Mourali MS, Addad F. Design and Rationale of the National Tunisian Registry of Heart Failure (NATURE-HF): Protocol for a Multicenter Registry Study. JMIR Res Protoc. 2021 Oct 27;10(10):e12262. doi: 10.2196/12262. PMID 34704958